CLINICAL TRIAL: NCT07393945
Title: Perioperative Human-Centered Communication on AI-Supported Real-Time Imaging and Its Effects on Preoperative Anxiety and Perceived Control: A Randomized Controlled Trial
Brief Title: Perioperative Human-Centered Communication on AI-Supported Real-Time Imaging
Acronym: XAI-COMM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Volkan Gokmen, Assistant Professor, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AI-XAI-RTI-PA-2026
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Preoperative Anxiety; Perceived Control
Keywords: Artificial intelligence; Explainable AI; Human-centered communication; Perioperative care; Real-time imaging; Randomized controlled trial

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either an intervention group receiving standard preoperative information plus a structured, human-centered explanation about AI-supported real-time imaging systems, or a control group receiving standard preoperative information alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human-Centered AI Communication (Experimental): Participants in this arm will receive standard preoperative information plus a structured, human-centered, non-technical explanation about AI-supported real-time imaging systems, focusing on their role, limitations, and relevance to patient safety.
  Interventions: Behavioral: Human-Centered Explainable AI Communication
- Standard Preoperative Information (Active Comparator): Participants in this arm will receive standard preoperative information routinely provided by the institution, without additional information related to AI-supported real-time imaging systems.
  Interventions: Other: Standard Preoperative Information

INTERVENTIONS:
Behavioral: Human-Centered Explainable AI Communication — A brief (approximately 5-7 minutes), face-to-face, structured communication delivered by a nurse, providing a non-technical and patient-centered explanation of AI-supported real-time imaging systems, including their general purpose, limitations, and relationship to patient safety. No AI software, device, or imaging system is tested or evaluated as part of the intervention.
  Arms: Human-Centered AI Communication
Other: Standard Preoperative Information — Routine preoperative information provided by the institution as part of standard clinical care.
  Arms: Standard Preoperative Information

SUMMARY:
This study investigates whether a structured, human-centered explanation about the use of artificial intelligence (AI)-supported real-time imaging systems can reduce preoperative anxiety and improve patients' sense of control before elective surgery.

Advances in medical imaging and AI technologies have increased their visibility in clinical settings, including the perioperative period. However, limited information is available on how explanations about such technologies influence patients' psychological responses. In particular, uncertainty or misunderstanding about AI-supported systems may contribute to increased anxiety in some patients.

In this randomized controlled trial, adult patients scheduled for elective surgery will be assigned to one of two groups. The control group will receive standard preoperative information routinely provided by the hospital. The intervention group will receive standard information plus a short, structured, and non-technical explanation about AI-supported real-time imaging systems, focusing on their role, limitations, and relevance to patient safety.

Levels of preoperative anxiety and perceived control will be assessed before and after the information session using validated questionnaires. The study does not test or evaluate the technical performance of any AI system. Instead, it focuses on how communication and explanation about AI-supported technologies may influence patients' psychological preparedness for surgery.

The findings may help inform human-centered and ethically responsible approaches to communicating about advanced technologies in perioperative care.

DETAILED DESCRIPTION:
The increasing integration of artificial intelligence (AI)-supported real-time imaging systems into clinical workflows has transformed diagnostic and perioperative practices. While the technical performance and clinical utility of these systems have been widely studied, considerably less attention has been given to how patients perceive and psychologically respond to information about AI-supported technologies used in their care.

Preoperative anxiety is a common psychological stressor among surgical patients and is associated with adverse perioperative outcomes, including increased postoperative pain, delayed recovery, and reduced patient satisfaction. Perceived control has been identified as a key psychological factor that can buffer the negative effects of anxiety, particularly in high-uncertainty clinical contexts such as the perioperative period.

This single-center, parallel-group randomized controlled trial is designed to evaluate the psychological effects of a structured, human-centered communication intervention related to AI-supported real-time imaging systems. Adult patients scheduled for elective surgery will be randomly assigned in a 1:1 ratio to either an intervention group or a control group following baseline assessment.

Participants in the control group will receive standard preoperative information routinely provided by the institution. Participants in the intervention group will receive standard information plus a brief (approximately 5-7 minutes), face-to-face, structured explanation about AI-supported real-time imaging systems. The intervention will use non-technical, patient-centered language and will address the general purpose of such systems, their role and limitations in clinical practice, and their relationship to patient safety and clinical decision-making. The intervention does not involve the use, testing, or evaluation of any specific AI software, device, or imaging system.

Preoperative anxiety and perceived control will be assessed at baseline (prior to randomization) and again after the information session, before surgery. The primary analyses will compare changes in anxiety and perceived control between the intervention and control groups, with baseline values accounted for in the statistical models.

This study does not aim to assess the diagnostic accuracy, technical performance, or clinical effectiveness of AI-supported imaging systems. Instead, it focuses on the communication and explanatory context surrounding such technologies, with the goal of informing human-centered, transparent, and ethically responsible strategies for integrating AI-supported systems into perioperative care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Scheduled for elective surgical procedures.
* Able to communicate in Turkish.
* At least primary school literacy.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Emergency surgical procedures.
* Known diagnosis of psychiatric disorders.
* Current use of anxiolytic or antidepressant medications.
* Cognitive impairment or communication barriers that may interfere with study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Change in Preoperative Anxiety Level | From baseline (before randomization) to immediately after the intervention and before surgery (approximately 10-15 minutes total).
  Preoperative anxiety will be assessed using the Amsterdam Preoperative Anxiety and Information Scale (APAIS).
  The primary outcome is the change in anxiety score between baseline (before randomization, T0) and after the intervention (prior to surgery, T1).
  Higher scores indicate higher levels of preoperative anxiety.

SECONDARY OUTCOMES:
Change in Perceived Control Level | From baseline (before randomization) to immediately after the intervention and before surgery (approximately 10-15 minutes total).
  Perceived control will be measured using a validated perceived control scale adapted for the healthcare setting.
  The secondary outcome is the change in perceived control score from baseline (T0) to after the intervention (T1), prior to surgery.
  Higher scores indicate a higher level of perceived control.

CONTACTS AND LOCATIONS:
Locations (1):
- Ağrı Training and Research Hospital, Ağrı, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the small sample size and the sensitive nature of psychological outcomes collected in this study.

REFERENCES:
- [Background] Chan SL, Sit JWH, Ang WW, Lau Y. Virtual reality-enhanced interventions on preoperative anxiety symptoms in adults undergoing elective surgery: A meta-analysis and meta-regression. Int J Nurs Stud. 2024 Dec;160:104886. doi: 10.1016/j.ijnurstu.2024.104886. Epub 2024 Aug 30. PMID 39270596
- [Background] Xu H, Hou J, Zhou J, Wang S. Effects of Virtual Reality on Preoperative Anxiety in Adult Patients: An Updated Meta-analysis. J Perianesth Nurs. 2025 Apr;40(2):422-430.e3. doi: 10.1016/j.jopan.2024.05.009. Epub 2024 Sep 26. PMID 39340515
- [Background] Guo P, East L, Arthur A. A preoperative education intervention to reduce anxiety and improve recovery among Chinese cardiac patients: a randomized controlled trial. Int J Nurs Stud. 2012 Feb;49(2):129-37. doi: 10.1016/j.ijnurstu.2011.08.008. Epub 2011 Sep 22. PMID 21943828
- [Background] Yahagi M, Hiruta R, Miyauchi C, Tanaka S, Taguchi A, Yaguchi Y. Comparison of Conventional Anesthesia Nurse Education and an Artificial Intelligence Chatbot (ChatGPT) Intervention on Preoperative Anxiety: A Randomized Controlled Trial. J Perianesth Nurs. 2024 Oct;39(5):767-771. doi: 10.1016/j.jopan.2023.12.005. Epub 2024 Mar 21. PMID 38520470